CLINICAL TRIAL: NCT04610216
Title: Investigation of the Automatic Technology on the Naída M Hearing Devices
Status: Completed | Type: Observational
Sponsor: Advanced Bionics AG (Industry)
Responsible Party: Sponsor
Other Study IDs: ABIntl-20-15
Record Dates: First submitted 2020-10-07; First posted 2020-10-30 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2021-03

CONDITIONS: Cochlear Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bilateral users: two implant systems: For bilateral CI users two Naida CI M sound processors (one per ear) will be used during the study.
  Interventions: Device: Naida CI M hearing device
- Bimodal users: hearing aid contralateral: For bimodal subjects there will be one Naida CI M sound processor on the implanted ear as well as one hearing aid on the contralateral ear.
  Interventions: Device: Naida CI M hearing device

INTERVENTIONS:
Device: Naida CI M hearing device — speech intelligibility measurement with Naida CI M hearing device

SUMMARY:
In this clinical trial, an un-controlled, repeated measures open design with within-subject comparison will be used to evaluate the effect of the device under investigation on sound perception. This design was shown to be successful in previous studies for the evaluation of sound coding strategies.

Furthermore, a within-subject comparison decreases the variance in the results allowing for fewer subjects when the population using the investigational device is not large in general.

DETAILED DESCRIPTION:
The primary endpoint of this clinical investigation is the difference in speech intelligibility measured in percent correct with AutoZoomControl compared to an omnidirectional microphone on Naída M hearing devices.The Naída CI M90 sound processor is a behind-the-ear (BTE) sound processor based on the Phonak Marvel hearing aid platform. It replaces the market approved Naída CI Q-Series processors. The Naída Link M90 hearing aid is a behind-the-ear (BTE) hearing aid based on the Phonak Marvel hearing aid platform. It is especially designed to be used for bimodal CI users equipped with a Naída CI M90 sound processor.

ELIGIBILITY:
Inclusion Criteria:

* · CI users with a CII, HiRes90K (Advantage) or HiRes Ultra (3D) implant system Bilateral users: two implant systems Bimodal users: hearing aid contralateral

  * Minimum of 18 years of age
  * Minimum of six months experience with their implant system
  * Minimum of six months experience with the Naída CI Q-Series sound processor
  * Ability to give feedback on sound quality
  * Speech reception thresholds of no more than 5 dB SNR > 10 at the French Matrix test obtained during previous visits in the clinical routine
  * Fluent in French language

Exclusion Criteria:

* Difficulties additional to hearing impairment that would interfere with the study procedures

  * Concurrent participation in other study
  * Incapacity for consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intended users of the Naída M hearing system are people who suffer from profound sensorineural hearing losses up to complete deafness. The users could be recipients that are already users of an Advanced Bionics CI but also people who suffer from deafness or profound hearing loss and were not previously equipped with a hearing device. In case of contralateral acoustic hearing, the user might use a Naída CI M90 on the side with profound sensorineural hearing loss and a Naída Link M90 as a hearing aid on the contralateral side to aid the residual acoustic hearing.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Difference in speech intelligibility in noise | 2 months
  The primary endpoint of this clinical investigation is the difference in speech intelligibility measured in percent correct with AutoZoomControl compared to an omnidirectional microphone on Naída M hearing devices. The French Matrix Test will be used and percentage correct will be recorded.

SECONDARY OUTCOMES:
Differences in speech perception in noise | 2 months
  ZoomControl versus Omnidirectional microphone and AutoZoomControl versus ZoomControlon Naída M hearing devices will be compared.
  The French Matrix Test will be used and percentage correct will be recorded.
Differences in localization abilities | 2 months
  AutoZoom control versus Omnidirectional microphone, ZoomControl versus Omnidirectional microphone and AutoZoomControl versus ZoomControlon Naída M hearing devices will be compared.
  The directions (0,+/-90,180 degrees) from where the sentences of the French Matrix Test are presented have to be determined.
  Percentage correct will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Angélica Pérez-Fornos, Dr, Principal Investigator — angelica.perez-fornos@hcuge.ch
Locations (1):
- Hôpitaux Universitaires de Genève (HUG), Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No